CLINICAL TRIAL: NCT06371989
Title: Vacuum Assisted Biopsy and Surgery Correlation in HER2 and TN Breast Cancer Subtypes MRI Responders After Neoadjuvant Therapy: BISUCO TRIAL
Acronym: BISUCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19/160
Record Dates: First submitted 2024-03-26; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Breast Biopsy
Keywords: Neoadjuvant response; Vacuum assisted biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Image-Guided Vacuum assisted biopsy of Tumor Site (Experimental): Image-guided biopsy of the tumor bed and coil area performed before surgery
  Interventions: Procedure: Image guided vacuum assisted biopsy

INTERVENTIONS:
Procedure: Image guided vacuum assisted biopsy — Image guided VAB of tumor site. A needle is inserted into the affected tumor bed area using an US or stereotactic method to collect cells or tissue from a tumor mass.

SUMMARY:
BACKGROUND AND CURRENT STATUS:

Advancements in neoadjuvant systemic treatments (NST) for HER2 positive and triple-negative (TN) breast cancer (BC) subtypes have led to high rates of pathologic complete response (pCR), raising questions about the necessity of subsequent surgery, especially for those undergoing adjuvant radiotherapy. While Magnetic Resonance Imaging (MRI) remains the most effective imaging technique for assessing neoadjuvant treatment response, surgery is still required to confirm pCR in cases of almost complete or complete MRI response (iCR). To safely avoid surgery in these BC "exceptional responders," a technique with high negative predictive value is imperative.

OBJECTIVE:

This study aims to establish the diagnostic efficacy of image-guided vacuum-assisted biopsy (VAB) in assessing pathological complete response (pCR) after NST in HER2 positive or TN breast cancer subtypes, particularly those showing post NST-MRI complete or almost complete response.

METHODS:

A prospective study was conducted at "Hospital Universitario 12 de Octubre de Madrid" from June 25, 2018, to October 25, 2029. Twenty-five patients with HER2-positive or TN operable invasive ductal carcinoma (IDC) BC subtype, at stages cT1-3/N0-2 undergoing primary NST and showing complete or almost complete response on post NST-MRI, were enrolled. Ultrasound or stereotactic-guided vacuum-assisted biopsy (VAB) of the previous clip and tumor bed area was performed before surgery. VAB pathological results were compared with surgical pathological results to evaluate the diagnostic efficacy of predicting pCR with VAB after NST. Pathological representativeness of the VAB sample was ensured. pCR was defined as the absence of invasive ductal carcinoma and in situ ductal carcinoma.

DETAILED DESCRIPTION:
BACKGROUND AND CURRENT STATUS:

Currently, advancements in neoadjuvant systemic treatments (NST) for HER2 and TN (triple-negative) breast cancer (BC) subtypes achieve high rates of pathologic complete response (pCR), prompting questions about the necessity of subsequent surgery, particularly for those undergoing adjuvant radiotherapy.

Although MRI (Magnetic Resonance Imaging) is the most effective imaging technique for assessing neoadjuvant treatment response we continue need to do surgery to confirm pcR in almost MRI imaging complete response (iCR) and iCR.

To safe avoiding surgery in this BC "exceptional responders" subtypes we need to find a high negative predictive value technique.

OBJECTIVE:

To establish the diagnostic efficacy of guided image vacuum-assisted biopsy (VAB) in assessing pathological complete response (pCR) after neoadjuvant systemic therapy (NST) in HER2 or Triple Negative (TN) breast cancer (BC) subtypes, showing post NST-MRI complete or almost complete response.

METHODS:

A prospective study was conducted at a tertiary university hospital from March 2019 to October 2023 25 patients with HER2-positive or TN operable invasive ductal carcinoma (IDC) BC subtypes, at stages cT1-3/N0-2 undergoing primary neoadjuvant systemic therapy (NST) and showing complete or almost complete response on post NST-MRI, were enrolled in the study.

A 7G ultrasound or stereotactic guided vacuum-assisted biopsy (VAB) was performed of the previous clip marked tumour bed area before the surgery.

Then a comparison of the VAB pathological results with the surgical pathological results to evaluate the diagnostic efficacy (validity and safety) of predicting residual carcinoma pathologic complete response (pCR) with VAB after NST was made.

Pathological representativeness of the VAB sample is mandatory including only the cases with post treatment changes and pathological correlation of the bed tumour area.

pCR was defined as the absence of invasive ductal carcinoma and in situ ductal carcinoma.

The study's hypothesis aims to achieve a VAB Negative Predictive Value (NPV) to detect residual carcinoma over 90%. Additionally, accuracy, sensitivity, positive predictive value, and specificity are calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Biopsy-proven operable breast IDC non-otherwise specified (no other subtypes) with or without DCIS
* HER2-positive (score 3+ in immunohistochemistry or HER2 amplification in FISH) or TN subtypes as per immunohistochemistry
* Stages cT1-2/N0-2/M0
* Administration of standard complete neoadjuvant systemic treatment
* Complete or almost complete response on breast post NST-MRI

Exclusion Criteria:

* Uncompleted NST or non-operable breast carcinoma
* Associated suspicious microcalcifications on diagnostic mammogram measuring more than 20mm
* Proven multicentric or multifocal disease
* High-risk patients
* Personal history of breast cancer (ipsilateral or contralateral)

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
The negative Predictive Value (NPV), Positive predictive value, specificity and sensibility of the VAB compared to Standard Surgery with Pathologic Evaluation | 15 days
  Ultrasound or stereotactic-guided vacuum-assisted biopsy (VAB) of the previous clip and tumor bed area was performed before surgery. VAB pathological results were compared with surgical pathological results to evaluate the NPV, PPV , specificity and sensibility of predicting pCR with VAB after NST

CONTACTS AND LOCATIONS:
Overall Officials: sara jimenez arranz, Principal Investigator — Hospital Universitario 12 de Octubre Madrid
Locations (1):
- Sara Jimenez Arranz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 months